CLINICAL TRIAL: NCT02230345
Title: Study of the Effects of a Probiotic Yoghourt on the Metabolic Health of Normal Male Volunteers
Brief Title: Effects of a Probiotics on the Health of Normal Young Males
Acronym: FFF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Collaborators: Agroscope Liebefeld-Posieux Research Station ALP (Other)
Responsible Party: Principal Investigator, Francois Pralong, Full professor and Head, Service of Endocrinology, Diabetology and Metabolism, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 392/13
Record Dates: First submitted 2014-07-21; First posted 2014-09-03 (Estimated); Last update posted 2015-08-21 (Estimated); Status verified 2015-08

CONDITIONS: Inflammation; Dyslipidemia
Keywords: Probiotic; Yoghourt; Inflammation; Metabolomics
MeSH Terms: conditions — Inflammation; Dyslipidemias | interventions — Milk

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotic yogurt (Experimental): Daily administration, during two weeks, of two probiotic yogurts (200 mL each)
  Interventions: Dietary Supplement: Probiotic yogurt
- Acidified milk (Active Comparator): Daily administration, over two consecutive weeks, of an isocaloric dose (compared to probiotics) of unfermented acidified milk
  Interventions: Dietary Supplement: Acidified milk

INTERVENTIONS:
Dietary Supplement: Probiotic yogurt — Probiotic yogurt (fermented milk with Lactobacillus delbrueckii subsp. bulgaricus and Streptococcus thermophilus- YoFlex FD-DVS YC-X11 Fr, with the addition of Lactobacillus rhamnosus GG (LGG)- Culture Collection, University of Göteborg, Sweden CCUG 34291).
  Other Names: LGG
  Arms: Probiotic yogurt
Dietary Supplement: Acidified milk — Milk will consist in an isocaloric supplement (compared to probiotic yogurt) of unfermented milk
  Other Names: Milk
  Arms: Acidified milk

SUMMARY:
The important role played by the GI tract microflora on the metabolic health of an individual are increasingly recognized. In this respect, the initial studies of Metchinkoff that suggested a role of fermented food (specifically yoghourts ) to modulate the gut microflora have evolved into the concept of "probiotics". Probiotics are living microorganisms that bring a benefit to the host when administered in sufficient quantity (WHO/FAO, 2001).

Here the investigators will study, in normal young male volunteers, the potential to modulate post-prandial metabolic and inflammatory responses by the administration of a yoghourt containing the probiotic Lactobacillus rhamnosus (LGG).

DETAILED DESCRIPTION:
This is a prospective, randomized, double-blind and cross-over study designed to evaluate the potential of a probiotic (Lactobacillus rhamnosus) to modulate the post prandial metabolic and inflammatory response of normale healthy individuals.

After a wash out period during which volunteers will have to follow a diet devoid of all milk or milk-derived products, they will receive, in random order, either a daily dose of the probiotic, or a daily dose of acidified milk (control) for a total of three consecutive weeks. At the end of each of these period, they will be submitted to a day of investigation, during which their metabolic and inflammatory profile will be studied following the ingestion of a standard test meal. The potential for the probiotic to modulate the metabolic and inflammatory parameters will be evaluated.

The test meal will provide 1004Kcal under the form of 45.4g proteins (17%), 69g total fatty acids (62%), and 52.6g glucids (21%) as previously published (Schwander et al, J Nut 2014).

ELIGIBILITY:
Inclusion Criteria:

* Normal male with normal BMI (18.5-25 kg/m2)
* non smoker
* stable physical activity

Exclusion Criteria:

* Food intolerance (ceoliac disease, lactose intolerance, food allergies)
* Particular regimen (vegetarian...)
* Chronic disease (any)
* Elevated blood pressure
* Regular drug treatment
* Antibiotics treatement in the preceding six months
* >4 hrs/week of physical activity

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2014-03; Primary Completion 2014-12 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Metabolomic analyses | 6 hours
  Kinetics of metabolomic changes in blood during the 6 hours after meal ingestion, in presence of yogurt or placebo

SECONDARY OUTCOMES:
Glucose | 6 hours
  Kinetics of glucose during the 6 hours after meal ingestion, in presence of yogurt or placebo
Insulin | 6 hours
  Kinetics of insulin during the 6 hours after meal ingestion, in presence of yogurt or placebo
Glucagon like polypeptide-1 | 6 hours
  Kinetics of GLP-1 during the 6 hours after meal ingestion, in presence of yogurt or placebo
Gastric inhibitory polypeptide | 6 hours
  Kinetics of GIP during the 6 hours after meal ingestion, in presence of yogurt or placebo
Total cholesterol | 6 hours
  Kinetics of total cholesterol during the 6 hours after meal ingestion, in presence of yogurt or placebo
LDL-cholesterol | 6 hours
  Kinetics of LDL-cholesterol during the 6 hours after meal ingestion, in presence of yogurt or placebo
HDL-cholesterol | 6 hours
  Kinetics of HDL-cholesterol during the 6 hours after meal ingestion, in presence of yogurt or placebo
Non esterified fatty acids | 6 hours
  Kinetics of NEFAs during the 6 hours after meal ingestion, in presence of yogurt or placebo
Triglycerides | 6 hours
  Kinetics of triglycerides during the 6 hours after meal ingestion, in presence of yogurt or placebo
Interleukin-6 | 6 hours
  Kinetics of IL-6 will be measured in blood of volunteers after the administration of yogurt or placebo
Chemokine CCK2 | 6 hours
  Kinetics of CCK2 will be measured in blood of volunteers after the administration of yogurt or placebo
Chemokine CCK5 | 6 hours
  Kinetics of CCK5 will be measured in blood of volunteers after the administration of yogurt or placebo
Tunour necrosis factor alpha | 6 hours
  Kinetics of TNF-a will be measured in blood of volunteers after the administration of yogurt or placebo
Lipo-poly-saccharide | 6 hours
  Kinetics of LPS will be measured in blood of volunteers after the administration of yogurt or placebo

OTHER OUTCOMES:
Transcriptomic analyses | 6 hours
  Kinetics of gene expression in white blood cells during the 6 hours after meal ingestion, in presence of yogurt or placebo

CONTACTS AND LOCATIONS:
Overall Officials: Francois P Pralong, MD, Principal Investigator — Centre Hospitalier Universitaire Vaudois
Locations (1):
- Clinical research center, Lausanne University hospital, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Derived] Vionnet N, Munger LH, Freiburghaus C, Burton KJ, Pimentel G, Pralong FP, Badertscher R, Vergeres G. Assessment of lactase activity in humans by measurement of galactitol and galactonate in serum and urine after milk intake. Am J Clin Nutr. 2019 Feb 1;109(2):470-477. doi: 10.1093/ajcn/nqy296. PMID 30721917
- [Derived] Pimentel G, Burton KJ, von Ah U, Butikofer U, Pralong FP, Vionnet N, Portmann R, Vergeres G. Metabolic Footprinting of Fermented Milk Consumption in Serum of Healthy Men. J Nutr. 2018 Jun 1;148(6):851-860. doi: 10.1093/jn/nxy053. PMID 29788433